CLINICAL TRIAL: NCT06053450
Title: The Effect of Essential Oil Inhalation Patches on Perceived Burn-out & Stress on an Inpatient Medical-surgery Unit.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Rachel G. Blier, Nurse Educator, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY02001908
Record Dates: First submitted 2023-08-10; First posted 2023-09-25 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-05

CONDITIONS: Nursing Personnel
Keywords: Essential Oil Inhalation Patches; Essential oil and nursing stress; Medical-Surgical unit

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Essential Oil Ptach (Experimental): The nursing staff will wear an essential oil patch for 2 weeks.
  Interventions: Other: Oil Inhalation Patch

INTERVENTIONS:
Other: Oil Inhalation Patch — Each participant will wear a patch for a work week (3 worked shifts) and then no patch is worn for a week. This alternates for a total of a month.
  Other Names: Quella; Elequil

SUMMARY:
The purpose of this clinical study is to compare the use of an essential oil inhalation patch in medical surgical nurses on perceived burn-out and stress.

The main question is can essential oil inhalation patches decrease perceived burn-out and stress.

Participants will

* Take part in the study over 30 days, alternating weeks, resulting in each participant using six patches over six shifts.
* Complete anonymous Perceived Stress Survey (PSS) before the study begins and at the conclusion of the study.
* Participants will also complete a (different) survey after two weeks.

DETAILED DESCRIPTION:
Essential Oil inhalation patches are a nonpharmacological option that is worn by the nursing staff on an inpatient medical-surgical unit to determine the efficacy of patch on staff perceived stress & burn-out levels. Each participant will wear a new patch during six work shifts. Location is on chest or the ID badge area where it can be easily accessed to. The patch provides up to 8 hours of aromatic support. The patches use a unique patented technology that slows the release of the aromatic molecules while maintaining the purity and vitality of the essential oil. The FDA approved medical adhesive patches are roughly 1x1" in size, and are inhalation only- no contact of essential oils on skin. The patch is portable and discreet. No overwhelming aroma for others. The patch has directions for use on package with an expiration date. Used for a non-specific purpose for stress reduction environment for this study.

ELIGIBILITY:
Inclusion Criteria:

* Full time employee (Nurse, LPN, or LNA) working on L3WD and L4WC
* At least 18 years of age

Exclusion Criteria:

* Pregnant/breastfeeding or planning to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2025-06-30 (Actual); Primary Completion 2025-11-20 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Change in baseline perceived stress as measured by the Perceived Stress Scale | 4 weeks
  Scores are measured on 0-4 scale with 0 indicating never and higher scores are more frequent.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel G. Blier, MSN,RN, Principal Investigator — DHMC
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spence Laschinger HK, Leiter MP. The impact of nursing work environments on patient safety outcomes: the mediating role of burnout/engagement. J Nurs Adm. 2006 May;36(5):259-67. doi: 10.1097/00005110-200605000-00019. PMID 16705307